CLINICAL TRIAL: NCT01342549
Title: Treatment Strategy for Alcohol Use Disorders in Veterans With TBI
Acronym: AUD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D7201-I
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-05

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Use Disorders; Traumatic Brain Injury; Mood and Anxiety Disorders
MeSH Terms: conditions — Alcoholism; Brain Injuries, Traumatic; Anxiety Disorders | interventions — Valproic Acid; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): sodium valproate
  Interventions: Drug: Valproate
- Arm 2 (Active Comparator): naltrexone
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Valproate — 250mg per day 30 minutes after a meal. Dosages will be increase as tolerated to a maximum recommended dosage of 60 mg per kg per day. Usual dosage is between 1250mg to 2000mg per day
  Other Names: Depakote ER
  Arms: Arm 1
Drug: Naltrexone — 25mg per day, taken by mouth for 7 days, then 50mg per day
  Other Names: Revia
  Arms: Arm 2

SUMMARY:
The purpose of this research study is to understand the effectiveness of valproate (a common mood stabilizer) to further reduce alcohol misuse when given in addition to attending an alcohol rehabilitation program as well as the treatment of mood disorders or PTSD. The main goal of this project is to understand if people receiving valproate will have a better recovery than people receiving the standard treatment for alcohol dependence: naltrexone.

DETAILED DESCRIPTION:
Veterans are vulnerable to develop complex forms of addictive disorders characterized by the presence of traumatic brain injury and psychiatric conditions such as post-traumatic stress disorder and mood disturbances. Alcohol use disorders are frequently observed among veterans and exert a detrimental effect on community reintegration after deployment. Attending to this veteran health problem, the VA is devoting extraordinary efforts to develop adequate treatment strategies. In this study we will evaluate treatment outcomes and identify specific factors that influence alcohol use disorders treatment response in a VA Intensive Outpatient Program offering rehabilitation treatment to the growing number of veterans with alcohol use disorders. Cooperation between researchers and clinical staff will allow optimizing treatment strategies that enhance the recovery of veterans with alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Veterans attending alcohol use disorders rehabilitation treatment within the VA
* Presence of a diagnosis of alcohol dependence according to DSM-IV
* A history of heavy drinking
* Absence of withdrawal symptoms

Exclusion Criteria:

* Evidence of other substance abuse different from nicotine or cannabis (DSM-IV criteria) or by 2 consecutive positive urine drug screens
* Unstable medical conditions such as severe heart disease, liver or renal failure or evidence of neoplasia.
* Liver Enzymes (ALT, AST) serum levels >3 times the upper limit of normal
* Unstable psychiatric conditions that requires treatment in a more structured setting (i.e. active SI, worsening psychotic symptoms or acute mania)
* Diagnosis of schizophrenia or schizoaffective disorder
* Requiring therapy with valproate or naltrexone or has a history of significant side effects from either study drug
* Requiring therapy with topiramate, lamotrigine or carbamazepine
* Requiring chronic treatment with opioid analgesics for refractory pain
* Failed 3 previous intensive alcohol rehabilitation programs in the past 2 years
* Females

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo E Jorge, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (2):
- United States (2):
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: sodium valproate
  Valproate: 250mg per day 30 minutes after a meal. Dosages will be increase as tolerated to a maximum recommended dosage of 60mg per day. Usual dosage is between 1250mg to 2000mg per day
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1. Veterans age 18 to 60 2. Presence of a diagnosis of alcohol dependence (DSM-IV criteria); 3. A recent history of heavy drinking defined as 5 or more drinks in a sitting at least twice in a week during the previous 2 months;4. Absence of withdrawal symptoms CIWA-Ar (94);5. Presence of a knowledgeable informant
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age range of 18-60. We decided to exclude patients over 60 years in order to avoid significant confounders such as the neurodegenerative changes associated with aging as well as those related to the presence of cerebrovascular pathology, a frequent complication observed among older veterans. 2. Presence of a diagnosis of alcohol dependence according to DSM-IV criteria.
  years | 46.71 (9.52) | 48.13 (8.79) | 47.42 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 31 | 31 | 62
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse to Heavy Drinking as Defined by Having 5 or More Drinks in a Sitting for Men and Will be Assessed Using the Time Line Follow Back for Recent Drinking Method. A Structured Questionnaire Will Review Alcohol Consumed on the Previous Week.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 31 | 31
Weeks | 8.78 (0.97) | 15.99 (1.36)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 12/31 | 10/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=31) | Arm 2 (N=31)
Drowsiness (Nervous system disorders) | 12 | 10
Nausea (Gastrointestinal disorders) | 3 | 9
Diarrhea (Gastrointestinal disorders) | 10 | 9
Sweating (Skin and subcutaneous tissue disorders) | 5 | 10
Abdominal Pain (Gastrointestinal disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes